CLINICAL TRIAL: NCT02038309
Title: Persistent Platelet Reactivity in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Dr Jean-Guillaume DILLINGER, Department of Cardiology, Hopital Lariboisière
Other Study IDs: PPRACS
Record Dates: First submitted 2014-01-12; First posted 2014-01-16 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2014-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; persistent platelet reactivity
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Study of persistent platelet reactivity during acute coronary syndrome. Patients are included at admission to the hospital. Platelet aggregation is evaluated by platelet function testing after blood sampling during hospitalization. No changes in treatment is planned.

DETAILED DESCRIPTION:
Blood samples are performed on day 2 and 4 and collected with usual blood samples and analyzed by the laboratory. Maximal aggregation intensity and velocity are measured by light transmission aggregometry induced by arachidonic acid (AA) or adenosine diphosphate (ADP). Platelet function analyzer will be also used. No changes in treatment in response to the results is planned.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome with elevation in troponin

Exclusion Criteria:

* anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
maximum aggregation intensity | day 2
  Light transmission aggregometry following exposition to arachidonic acid 0.5mg/ml during the acute phase (day2-day 5)

SECONDARY OUTCOMES:
Maximum aggregation intensity | Day 2
  Light transmission aggregometry following exposition to adenosine diphosphate during the acute phase (day2-day 5) and during the chronic phase (day 30-day 60)
Maximum aggregation intensity | Chronic phase (day 30 to day 60)
  Light transmission aggregometry following exposition to arachidonic acid 0.5mg/ml during the chronic phase (day 30-day 60)

OTHER OUTCOMES:
Major cardiovascular and cerebrovascular events (MACCE) | one year
  Major cardiovascular and cerebrovascular events : death, myocardial infarction, stroke, rehospitalisation and bleeding (academic research consortium) events at 1 year
microvascular resistance index | Day 1
  measurement during primary PCI on admission

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, MD-PhD, Study Director — Department of Cardiology - Lariboisiere Hospital - APHP
Locations (1):
- Department of Cardiology - Lariboisiere Hospital, Paris, France